CLINICAL TRIAL: NCT02208518
Title: Could Quantitative And Qualitative EUS-Elastography Results Be Affected By The Compression Rate And The Diameter Of The Region Of Interest (ROI)?
Brief Title: Quantitative And Qualitative Eus Elastography
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: ELASTOSONO-EUS1
Record Dates: First submitted 2014-03-04; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Normal Pancreatic Tissue
Keywords: Endoscopic Ultrasound elastography; Quantitative elastography; Qualitative elastography; Endoscopic Ultrasound; Elastography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Elastography analysis: Consecutive patients undergoing for upper endoscopy ultrasound
  Interventions: Procedure: endoscopy ultrasound elastography; Device: EUS-elastography

INTERVENTIONS:
Procedure: endoscopy ultrasound elastography — During a endoscopy ultrasound (EUS) procedure, in patients with normal pancreas at EUS, elastography was performed using a software already included in Hitachi-Avius machine, pressing the button and obtaining colors and pressure curve given by the software
Device: EUS-elastography

SUMMARY:
Endoscopic ultrasonography is considered the most accurate methods for the diagnosis and staging of chronic inflammatory and neoplastic pancreatic diseases. Differential diagnosis of solid pancreatic masses, however, remains a challenge and endoscopic ultrasound-guided fine needle aspiration is necessary. Recently, Endoscopic ultrasound elastography has been introduced as an alternative method to evaluate tissue stiffness of solid pancreatic masses, being an index of tissue elasticity, which may be related to histopathology features (hard tissue = blue = neoplastic and soft tissue = red-yellow-green = non-neoplastic). However, recently publications show different results using elastography. Moreover, a lack of data in Endoscopic ultrasound-elastography exist regarding the compression rate of the probe and the diameter of the region of interest under analysis in previously studies that by physics could affect the tissue elasticity.

Based on the hypothesis that elastography could be affected by compression rate of the probe and the diameter of the region of interest analyzed the present study aimed to evaluate the quantitative (strain ratio) and qualitative endoscopic ultrasound-elastography results determined by the compression rate of the probe (measured by the curve of compression in the second generation of elastography) and the diameter of the region of interest in normal pancreatic tissue.

DETAILED DESCRIPTION:
prospective study performed in patients undergoing for upper-endoscopic ultrasound from October 31-to end of November 2013. Endoscopic ultrasound-elastography was performed using linear Pentax-EUS and "Hitachi-Avius". The quantitative-strain ratio and qualitative endoscopic ultrasound-elastography was measured in the body of the pancreas taking in consideration the curve of the compression rate of the probe high: +0.4, middle: 0, low: -0.4 in the largest and smaller region of interest diameters. Analysis for qualitative elastography was obtained by the predominant color of the pancreatic area studied. Pictures where recorded and quantitative strain ratio data were calculated comparing endoscopic ultrasound-elastography of pancreatic tissue with soft tissue (normal mucosal layer: red). Finally, a comparative analysis was performed between the results with the mean normal value for quantitative strain ratio previously published for normal pancreatic tissue, and between the different compression rates of the probe.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic Ultrasound for evaluate submucosal tumors

Exclusion Criteria:

* age<18 or > 55; pregnancy
* history of: pancreatic disease
* choledocolithiasis
* symptoms of maldigestion
* alcohol abuse
* increased serum levels of pancreatic enzymes
* smokers
* Endoscopic Ultrasound with signs of chronic pancreatitis (Rosemont classification)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: primary care clinic: patients with upper gastrointestinal submucosal tumors for evaluation by endoscopic ultrasound
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Quantitative Strain Ratio and qualitative Color endoscopy ultrasound elastography | two months
  The quantitative Strain Ratio and qualitative Color endoscopy ultrasound elastography was measured in the normal body of the pancreas taking in consideration the curve of the compression rate probe high: +0.4 , middle: 0: less than +0.4 and more than -0.4 [around baseline=0], and low: -0.4 in the largest and smaller region of interest diameters. Analysis for qualitative color elastography was obtained by the predominant color of the pancreatic area studied. Pictures where recorded and quantitative strain ratio data were calculated comparing endoscopic ultrasound elastography of pancreatic tissue with soft tissue (normal mucosal layer: red).

OTHER OUTCOMES:
Highest compression rate of the probe | 4 weeks
  the curve of the Highest compression rate of the probe: +0.4 , in the largest and smaller region of interest diameters
Middle compression rate of the probe | 4 weeks
  the curve of the Middle compression rate of the probe: 0: less than +0.4 and more than -0.4 [around baseline=0], in the largest and smaller region of interest diameters.
Lower compression rate of the probe | 4 weeks
  the curve of the Lower compression rate of the probe: -0.4 in the largest and smaller region of interest diameters
Qualitative elastography | 8 weeks
  Analysis for qualitative elastography was obtained by the predominant color of the pancreatic area studied.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD, Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas, Guayaquil, Guayas, Ecuador

REFERENCES:
- [Result] Iglesias Garcia JJ, Larino Noia J, Alvarez Castro A, Cigarran B, Dominguez Munoz JE. Second-generation endoscopic ultrasound elastography in the differential diagnosis of solid pancreatic masses. Pancreatic cancer vs. inflammatory mass in chronic pancreatitis. Rev Esp Enferm Dig. 2009 Oct;101(10):723-30. doi: 10.4321/s1130-01082009001000009. English, Spanish. PMID 19899942
- [Result] Iglesias-Garcia J, Larino-Noia J, Abdulkader I, Forteza J, Dominguez-Munoz JE. Quantitative endoscopic ultrasound elastography: an accurate method for the differentiation of solid pancreatic masses. Gastroenterology. 2010 Oct;139(4):1172-80. doi: 10.1053/j.gastro.2010.06.059. Epub 2010 Jun 27. PMID 20600020
- [Result] Dawwas MF, Taha H, Leeds JS, Nayar MK, Oppong KW. Diagnostic accuracy of quantitative EUS elastography for discriminating malignant from benign solid pancreatic masses: a prospective, single-center study. Gastrointest Endosc. 2012 Nov;76(5):953-61. doi: 10.1016/j.gie.2012.05.034. Epub 2012 Jul 31. PMID 22854060
- [Result] Giovannini M, Hookey LC, Bories E, Pesenti C, Monges G, Delpero JR. Endoscopic ultrasound elastography: the first step towards virtual biopsy? Preliminary results in 49 patients. Endoscopy. 2006 Apr;38(4):344-8. doi: 10.1055/s-2006-925158. PMID 16680632